CLINICAL TRIAL: NCT01378572
Title: Electrophysiologic and Morphologic Assessment of the Substrate to Guide Implantation of Defibrillators in Dilated Cardiomyopathy
Acronym: EMOSIDD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Texas Cardiac Arrhythmia Research Foundation (Other); Cardiac Arrhythmia Research Center, Centro Cardiologico Monzino, Milan, Italy (Unknown); Policlinico Casilino ASL RMB, Rome, Italy (Unknown); Dell'Angelo Hospital, Mestre-Venice, Italy (Unknown)
Responsible Party: Andrea Natale, Texas Cardiac Arrhythmia Institute, St David's Medical Center, Austin, TX, USA
Other Study IDs: SDMC060911
Record Dates: First submitted 2011-06-21; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Dilated Cardiomyopathy; Primary Prevention of Sudden Cardiac Death; Implantable Cardioverter Defibrillator
Keywords: ICD; sudden cardiac death; mapping
MeSH Terms: conditions — Cardiomyopathy, Dilated; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
With the present study the investigators intend to identify the morphologic and electrophysiologic substrate markers of increased arrhythmic risk in patients with dilated cardiomyopathy undergoing implantation of a defibrillator for the primary prevention of sudden cardiac death. Moreover, the investigators also aim to identify if there is any electrophysiological substrate modification at the time of the first arrhythmic event in these patients. To this aim, the investigators will prospectively correlate electroanatomic mapping and cardiac magnetic resonance findings with arrhythmic events, in order to identify substrate markers of increased arrhythmic risk in patients with dilated cardiomyopathy, who are therefore more likely to benefit from a defibrillator implantation. Furthermore, electroanatomic mapping will be repeated at the time of the first arrhythmic event and compared with that at baseline, in order to evaluate any electrophysiological substrate changes.

DETAILED DESCRIPTION:
A correct identification of patients at high risk of sudden cardiac death is crucial for a rational clinical management, since the demonstrated effectiveness of implantable cardioverter-defibrillators on the reduction of sudden cardiac death. Basing on the results of multiple clinical trials, left ventricular systolic function, measured as ejection fraction, is currently the only recommended tool to identify patients at higher risk of sudden death that would benefit from a prophylactic defibrillator. However, the systematic implementation of current recommendations results in a substantial number of inappropriate defibrillator implantations, while failing to prevent the majority of sudden deaths occurring in the general population. Unfortunately, at present time we have no other way to identify patients at higher risk of sudden cardiac death, since other proposed risk markers have not been consistently demonstrated of incremental value. Recent data suggest that several substrate markers, either assessed morphologically with magnetic resonance imaging, or electrophysiologically with invasive mapping procedures, may be helpful to identify subgroup of patients at higher arrhythmic risk. However, previous studies have been largely conducted on few patients, most were retrospective or with short follow-up.

We will submit patients with dilated cardiomyopathy undergoing implant of an implantable cardioverter defibrillator to a morphologic and electrophysiologic substrate evaluation including cardiac magnetic resonance with gadolinium contrast-enhancement study, and electroanatomic mapping with bipolar electrogram voltage and morphological analysis. The electroanatomic mapping and cardiac magnetic resonance will be repeated at the time of the first arrhythmic event.

We expect to define the role of anatomical and electrophysiological substrate abnormalities in determining malignant ventricular arrhythmias in patients with dilated cardiomyopathy, thus allowing a better risk stratification and prevention of sudden death.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 year-old with full capacity.
2. A New York Heart Association (NYHA) class II or III chronic, stable congestive heart failure (CHF).
3. A left ventricular ejection fraction (LVEF) of no more than 35 percent.

Exclusion Criteria:

1. Age <18 years or diminished capacity.
2. Patients with LVEF ≥ 35% or asymptomatic left ventricular dysfunction.
3. Patients with NYHA class IV CHF.
4. Patients with history of ventricular arrhythmias causing pre-syncope or syncope, cardiac arrest or a spontaneous episode of sustained ventricular tachycardia (VT) (≥30 seconds at rates of >100 bpm), unless these occurred within 48 hours of a myocardial infarction.
5. Females who are pregnant or have childbearing potential and are not using reliable methods of contraception.
6. Patients with history of restrictive, infiltrative, or hypertrophic cardiomyopathy; arrhythmogenic cardiomyopathy; constrictive pericarditis; congenital heart disease; surgically correctable valvular disease; and/or inoperable obstructive valvular disease.
7. Patients with reversible nonischemic cardiomyopathy such as acute viral myocarditis, alcohol-induced cardiomyopathy, peripartum cardiomyopathy, Takotsubo cardiomyopathy.
8. Patients with mechanical or biologic prosthetic cardiac valves.
9. Patients with history of a major psychiatric disorder, active alcohol/drug abuse, or noncompliance.
10. Coronary artery bypass graft surgery or percutaneous coronary intervention (balloon and/or stent angioplasty) within the past 90 days prior to enrollment.
11. Myocardial infarction within the past 90 days prior to enrollment.
12. Angiographic evidence of coronary disease sufficient to be a candidate for coronary revascularization and likely to undergo coronary artery bypass graft surgery and/or percutaneous coronary intervention and likely to undergo such a procedure in the foreseeable future.
13. Presence of any disease, other than the patient's cardiac disease, associated with a reduced likelihood of survival for the duration of the study, including but not limited to cancer, uremia (blood urea nitrogen >70 mg/dl or creatinine >3.0 mg/dl), respiratory failure, hepatic failure, etc.
14. Contraindication to cardiac magnetic resonance evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dilated cardiomyopathy (NYHA II-III heart failure, left ventricular ejection fraction <=35%) undergoing prophylactic ICD implantation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-11

PRIMARY OUTCOMES:
Arrhythmic Event | 2 years
  ICD shock on rapid sustained ventricular tachycardia or ventricular fibrillation or effective antitachycardia pacing.
Change in Arrhythmogenic Substrate | 2 years
  Change in the arrhythmogenic substrate in patients who will experience an arrhythmic event compared to a matched control group who will remain free from arrhythmic event.

SECONDARY OUTCOMES:
Heart failure events | 2 years
  Hospitalization for heart failure events
Death | 2 years
  All-cause mortality

CONTACTS AND LOCATIONS:
Locations (3):
- Texas Cardiac Arrhythmia Institute, St. David's Medical Center, Austin, Texas, United States
- Italy (2):
  - Centro Cardiologico Monzino, Milan
  - Policlinico "A. Gemelli", Rome